CLINICAL TRIAL: NCT02572089
Title: Phase 1, Pharmacokinetic Evaluation of Intranasal and Intramuscular Naloxone in Healthy Volunteers
Brief Title: Pharmacokinetic Evaluation of Intranasal and Intramuscular Naloxone in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Vince & Associates Clinical Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Naloxone-Phase1a-002
Record Dates: First submitted 2015-10-05; First posted 2015-10-08 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2015-10

CONDITIONS: Drug Overdose; Opioid-Related Disorders
MeSH Terms: conditions — Drug Overdose; Opioid-Related Disorders | interventions — Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 2mg Intranasal Naloxone (Experimental): Administer 0.1mL spray of the 20 mg/mL formulation in one nostril
  Interventions: Drug: Naloxone
- 4mg(a) Intranasal Naloxone (Experimental): Administer 0.1mL spray of the 20 mg/mL formulation in both nostrils
  Interventions: Drug: Naloxone
- 4mg(b) Intranasal Naloxone (Experimental): Administer 0.1mL spray of the 40mg/mL formulation in one nostril
  Interventions: Drug: Naloxone
- 8mg Intranasal Naloxone (Experimental): Administer 0.1mL spray of the 40mg/mL formulation in both nostrils
  Interventions: Drug: Naloxone
- Intramuscular Naloxone (Experimental): Administer 1mL of 0.4mg/mL formulation intramuscularly
  Interventions: Drug: Naloxone

INTERVENTIONS:
Drug: Naloxone

SUMMARY:
To determine the pharmacokinetics of 4 intranasal doses of naloxone compared to a 0.4 mg dose of naloxone administrated intramuscular and to identify an appropriate intranasal dose that could achieve systemic exposure comparable to an approved parenteral dose. To also determine the pharmacokinetics of two different concentrations of intranasal naloxone and finally, to determine the safety of intranasal naloxone with respect to nasal irritation.

ELIGIBILITY:
Inclusion Criteria:

* Be able to provide written consent
* Must have a BMI ranging from 18 to 30kg/m2, inclusive
* Must have adequate venous access
* Must not have any clinically significant concurrent medical conditions determine by medical history, physical examination, vital signs, and 12-lead electrocardiogram.
* Must agree to use a reliable double-barrier method of birth control from the start of screening until one week after completing the study. Oral contraceptives are prohibited.
* Must agree to not ingest alcohol, drinks containing xanthine greater than 500 mg/day (e.g., Coca Cola, coffee, tea, etc.), or grapefruit/grapefruit juice or participate in strenuous exercise 72 hours prior to admission through the last blood draw of the study.

Exclusion Criteria:

* Please contact clinical site directly for more information

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 720 minutes
  Measurement of serum naloxone prior to dosing and at times 2.5, 5, 10, 15, 20, 30, 45, 60, 120, 180, 240, 300, 360, 480 and 720 minutes after naloxone administration.
Time at Maximum Plasma Concentration (Tmax) | 720 minutes
  Measurement of serum naloxone prior to dosing and at times 2.5, 5, 10, 15, 20, 30, 45, 60, 120, 180, 240, 300, 360, 480 and 720 minutes after naloxone administration
Area Under the Concentration (AUC 0-t) | 720 minutes
  Time curve from time zero to last measurable concentration. Measurement of serum naloxone prior to dosing and at times 2.5, 5, 10, 15, 20, 30, 45, 60, 120, 180, 240, 300, 360, 480 and 720 minutes after naloxone administration
Area Under Curve (AUC 0-inf) | 720 minutes
  Time curve from time zero to infinity. Measurement of serum naloxone prior to dosing and at times 2.5, 5, 10, 15, 20, 30, 45, 60, 120, 180, 240, 300, 360, 480 and 720 minutes after naloxone administration
Half-life | 720 minutes
  The apparent terminal exponential half-life. Measurement of serum naloxone prior to dosing and at times 2.5, 5, 10, 15, 20, 30, 45, 60, 120, 180, 240, 300, 360, 480 and 720 minutes after naloxone administration

SECONDARY OUTCOMES:
Adverse events | minimum of 18 days
  will be reported from the start of the first session to the follow-up visit
Vital Signs | 480 minutes
  Measured at pre-dose and at times 30 , 60, 120 and 480 minutes after naloxone administration.
12-lead electrocardiogram | 480 minutes
  Measured at pre-dose and at times 60 and 480 minutes after naloxone administration.
Nasal Irritation Scoring | 24 hours
  Measured at pre-dose and at times 5, 30 , 60, 240 minutes and 24 hours after nasal naloxone administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Vince Associates Clinical Research, Overland Park, Kansas, United States